CLINICAL TRIAL: NCT05513430
Title: Pharmacological and Nonpharmacological Factors That Contribute Blood Pressure Control
Status: Completed | Type: Observational
Sponsor: Maltepe University (Other)
Collaborators: Istanbul University (Other)
Responsible Party: Principal Investigator, Asst. Prof. Zeynep Gunes Ozunal, M.D., Asst Prof, Maltepe University
Other Study IDs: 000001
Record Dates: First submitted 2017-08-24; First posted 2022-08-24 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Hypertension,Essential
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- controlled hypertension: Controlled hypertension was defined as systolic blood pressure (SBP) ≤139 mmHg and/or diastolic blood pressure (DBP)≤89 mmHg for non-diabetic patients, and as SBP ≤139 mmHg and/or DBP ≤84 mmHg for diabetic patients, based on the European Society of Hypertension (ESH) and of the European Society of Cardiology (ESC) guidelines. observational study
- uncontrolled hypertensive patients.: Individuals who had blood pressure levels above these values were defined as uncontrolled hypertensive patients.

SUMMARY:
Study is an observational study among hypertensive patients

DETAILED DESCRIPTION:
Objective: To investigate drug adherence and lifestyle behaviors affecting the blood pressure (BP) control among hypertensive patients that have uncontrolled and controlled BP.

ELIGIBILITY:
Patient inclusion criteria were as follows:

* aged between 38 and 74 years,
* hypertension diagnosis history of at least 6 months
* use of at least one antihypertensive medication.

Exclusion Criteria:

-not willing to join the clinical trial

Max Age: 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: hypertensive patients
Sampling Method: Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2014-06-16 (Actual); Primary Completion 2014-11-30 (Actual); Study Completion 2014-11-30 (Actual)

PRIMARY OUTCOMES:
health related quality of life. | at the time of the beginning of the study
  EQ-5D-3L turkish validation test
Age | at the time of the beginning of the study
  years
Gender | at the time of the beginning of the study
  Female/Male
BMI | at the time of the beginning of the study
  (kg/m2)

SECONDARY OUTCOMES:
complementary and alternative medicine use | at the time of the beginning of the study
  subjective reports from patients (yes/no)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mancia G, Fagard R, Narkiewicz K, Redon J, Zanchetti A, Bohm M, Christiaens T, Cifkova R, De Backer G, Dominiczak A, Galderisi M, Grobbee DE, Jaarsma T, Kirchhof P, Kjeldsen SE, Laurent S, Manolis AJ, Nilsson PM, Ruilope LM, Schmieder RE, Sirnes PA, Sleight P, Viigimaa M, Waeber B, Zannad F; Task Force Members. 2013 ESH/ESC Guidelines for the management of arterial hypertension: the Task Force for the management of arterial hypertension of the European Society of Hypertension (ESH) and of the European Society of Cardiology (ESC). J Hypertens. 2013 Jul;31(7):1281-357. doi: 10.1097/01.hjh.0000431740.32696.cc. No abstract available. PMID 23817082
- [Result] Özünal, Z. G., Tahirbegolli, I. A., Baykal, M., Belen, A. T. E. Ş., Tahirbegolli, B., KILIÇ, Y., ... & Üresin, A. Y. (2019). The drug adherence and lifestyle factors that contribute to blood pressure control among hypertensive patients.